CLINICAL TRIAL: NCT05962515
Title: Evaluation of the Efficacy of Ultrasound-Guided Dry Needling Therapy and Exercise Programme in Piriformis Muscle Syndrome
Brief Title: Efficacy of Ultrasound-Guided Dry Needling Therapy and Exercise in Piriformis Muscle Syndrome
Status: Completed | Type: Observational
Sponsor: Tepecik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, derya guner, Pain Physician, MD, Tepecik Training and Research Hospital
Other Study IDs: 2022/2/1
Record Dates: First submitted 2023-07-17; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Piriformis Muscle Syndrome; Dry Needling; Ultrasonography; Ultrasound Guided Dry Needling; Exercise Treatment
Keywords: piriformis muscle syndrome; pain; dry needling; exercise; ultrasound; neuralgia; interventional ultrasonography; physical therapy modalities
MeSH Terms: conditions — Piriformis Muscle Syndrome; Pain; Motor Activity; Neuralgia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: All patients in group 1 (n:22) had DN treatment applied to the piriformis muscle once a week for a total of 3 times under US guidance.
  Interventions: Procedure: ultrasound guided dry needling
- 2: All patients in group 2(n:22) had exercise programme for 3 weeks.
  Interventions: Procedure: ultrasound guided dry needling

INTERVENTIONS:
Procedure: ultrasound guided dry needling — Dry needling was applied in the intervention room with sterile conditions the patient in the prone position.The low frequency (2-5 MHz) transducer is placed in the gluteal region in a slightly oblique position and sonographic scanning is started. First, the large mountain shadow of the iliac crest and gluteus maximus muscle is sonographically visualized in the midline. Then the transducer is shifted inferiorly until the sciatic notch is visualized. When the sciatic notch, sciatic nerve and the pear-shaped piriformis muscle above it are visualized, the patient's knee is flexed and the leg is rotated internally and externally, and the typical sliding motion of the piriformis muscle is observed. After the target point is determined, a 22 G spinal needle is applied from lateral to medial or from medial to lateral with in plane technique. The needle is inserted and withdrawn several times until the switch response in the piriformis muscle is observed and extinguished
  Other Names: exercise programme

SUMMARY:
Piriformis muscle syndrome (PMS) is a neuromuscular disorder that can cause symptoms of hip joint motion limitation, buttock pain and tenderness, and numbness radiating to the back of the thigh due to compression or irritation of the sciatic nerve.In the etiology of PMS myofascial trigger points are the most common cause and also hypertrophy in the piriformis muscle tissue, inflammation, trauma, anatomical variations of the piriformis muscle or sciatic nerve may also cause the development of PMS . Physical examination supports the diagnosis of PMS and may help to eliminating competing diagnoses. Multiple physical examination maneuvers have been identified to help diagnose but no physical examination maneuver is diagnostic for PMS. Compression and deep palpation may also exacerbate buttock or gluteal pain. Electrodiagnostic tests are usually normal in FMS and useful in excluding other conditions such as lumbosacral radiculopathy .There is no gold standard treatment option for PMS, conservative treatment and lifestyle changes remain the mainstays for the treatment. Piriformis muscle stretching is the form of an exercise technique in physiotherapy method that is generally used for those patients. The exercises focused on relaxing the priformis muscle to increase the resting length of the muscle and reduce the potential sciatic nerve compression because of this thigtness. Dry needling (DN) therapy is a treatment method where myofascial trigger points are stimulated using acupuncture needles or injection needles .DN can be applied according to the anatomical landmark method or under the guidance of ultrasound (US) and fluoroscopic imaging. US guidance is important in the management of PMS, which allows imaging of specific deep muscle groups and avoids complications such as procedural pain and damage of neurovascular structures . There are no randomized controlled studies other than case series on the use and frequency of application of the US-guided DN technique in PMS. The aim of this study is to compare the effectiveness of dry needling treatment applied to the piriformis muscle once a week for a total of 3 times under US guidance and 3-week exercise program treatment in PMS. The secondary outcomes of this study is to evaluate and compare the effect of these treatment modalities on Visuel Analg Scale (VAS) scores ,Oswestry Disability Index (ODI), lower extremity functional scale (LEFS) and (Douleur Neuropathique 4 Questionare ) DN4 scores in PMS patients at 3 months follow up.

DETAILED DESCRIPTION:
In this observational study, between January 2022 and April 2023, after excluding other hip, lumbar, sacroiliac region and lower extremity pain etiology diagnoses, 44 patients aged 18-70 years who are clinically diagnosed with PMS are planned to be included in the study. The diagnosis is based on patient's history and physical examination, bearing positive FAIR test and/or tenderness or trigger point at the priformis muscle area and/or revealing the pain with maneuvers; such as Freiberg's maneuver , Beatty's maneuver and Pace's maneuver . The demographic data (age, sex, occupation, body mass index scores), the side of the pain will be noted. Each patient in the study will receive and sign an informed consent form.The patients will divide into two groups ; group 1 (n:22)will have DN treatment to the piriformis muscle once a week for a total of 3 times under US guidance, all patients in group 2 (n:22) will have exercise programme for 3 weeks. Overall pain severity will measure by using visual analogue scale (VAS). Pain disability will assess with the Oswestry Disability Index (ODI) questionnaire, Physical function will rate with Lower Extremity Functional Scale (LEFS). Presence and severity of neuropathic pain will evaluate according to Douleur Neuropathique 4 questionnare (DN4). To identify the outcomes of the treatment modalities, pre-treatment, post-treatment 1st month and 3th-month scores will be used. Patients with comorbidities that prevented interventional treatment (e.g., inflammatory diseases, uncontrolled diabetes mellitus, uncontrolled hypertension, malignancy, pregnancy, and severe psychiatric disorders), patients with other diagnoses that may cause hip and leg pain (e.g.,lumbar disc herniation, sciatic nerve injury history, sacroiliac and hip joint pathologies) those aged under 18 years old and patients who did not accept interventional or physical therapy modalities are going to exclude from the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with isolated Piriformis Muscle Syndrome
* The diagnosis is based on patient's history and physical examination, bearing positive FAIR (flexion, adduction, internal rotation) test and/or tenderness or trigger point at the priformis muscle area and/or revealing the pain with maneuvers; such as Freiberg's maneuver (forceful internal rotation of the extended thigh in the supine position), Beatty's maneuver (actively abducting the affected thigh in the lateral decubitus position) and Pace's maneuver (resisted abduction of both thighs in the seated position).

Exclusion Criteria:

* Patients with comorbidities that prevented interventional treatment (e.g., inflammatory diseases, uncontrolled diabetes mellitus, uncontrolled hypertension, malignancy, pregnancy, and severe psychiatric disorders),
* Patients with other diagnoses that may cause hip and leg pain (e.g.,lumbar disc herniation, sciatic nerve injury history, sacroiliac and hip joint pathologies)
* Aged under 18 years old
* Patients who will not accept interventional or physical therapy modalities

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients were divided into two groups as those who will accept DN treatment (Group 1 -n: 22) and those who will have physical exercise treatment (Group 2- n: 22). All patients in group 1 will have DN treatment to the piriformis muscle once a week for a total of 3 times under US guidance.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Visuel Analogue Scale | change from baseline VAS scores at 3 months
  Overall pain severity was measured by using a 0 to 100 mm scale visual analogue scale (VAS).

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) questionnaire, | change from baseline ODI scores at 3 months
  Oswestry Disability Index (ODI) questionnaire, which measures pain disability consists of ten questions, each with six options . The questions include the pain intensity, ability to work, perform self care, sit ,stand, travel, lift, sleep pattern, socializing and sexual life. Every question was scored between 0 and 5 points. The highest score is 50 if all questions were answered, and indicates severe disability for the participant.
lower extremity functional scale (LEFS) | change from baseline LEFS scores at 3 months
  The LEFS consists of 20 items to rate the ability of functional status in performing different physical activities due to musculoskeletal problems affecting the lower extremities. Each question has five point scale, from 0 to 4 (0: unable to do the activity, 1: quite, 2: moderate, 3: somewhat, 4: no difficulty). The total score ranges from 0 to 80, with higher scores indicate better functional status
Douleur Neuropathique 4 questionnare (DN4) | change from baseline DN4 scores at 3 months
  The questionnaire derived from this list, called DN4, included a series of four questions consisting of both sensory descriptors and signs related to bedside sensory examination. This provisional questionnaire was not intended to be exhaustive and was deliberately restricted to a minimum of simple and presumably discriminant items requiring yes or no responses.

CONTACTS AND LOCATIONS:
Locations (1):
- Tepecik Training and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tabatabaiee A, Takamjani IE, Sarrafzadeh J, Salehi R, Ahmadi M. Ultrasound-guided dry needling decreases pain in patients with piriformis syndrome. Muscle Nerve. 2019 Nov;60(5):558-565. doi: 10.1002/mus.26671. Epub 2019 Aug 27. PMID 31415092
- [Result] Fusco P, Di Carlo S, Scimia P, Degan G, Petrucci E, Marinangeli F. Ultrasound-guided Dry Needling Treatment of Myofascial Trigger Points for Piriformis Syndrome Management: A Case Series. J Chiropr Med. 2018 Sep;17(3):198-200. doi: 10.1016/j.jcm.2018.04.002. Epub 2018 Aug 26. PMID 30228811
- [Result] Misirlioglu TO, Akgun K, Palamar D, Erden MG, Erbilir T. Piriformis syndrome: comparison of the effectiveness of local anesthetic and corticosteroid injections: a double-blinded, randomized controlled study. Pain Physician. 2015 Mar-Apr;18(2):163-71. PMID 25794202